CLINICAL TRIAL: NCT06043362
Title: Randomized Placebo-controlled Trial of Nicotine Pouches in Smokers
Brief Title: Use of Nicotine Pouches Among Daily Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jonathan Foulds, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00023056; 1U54DA058271 (NIH)
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 0 mg + Smooth flavor (Experimental): Participants are provided with zero strength (0 mg) nicotine pouches with smooth flavor.
  Interventions: Other: 0 mg nicotine pouch; Other: Smooth nicotine pouch
- 3 mg + Smooth flavor (Experimental): Participants are provided with medium strength (3 mg) nicotine pouches with smooth flavor.
  Interventions: Other: 3 mg nicotine pouch; Other: Smooth nicotine pouch
- 6 mg + Smooth flavor (Experimental): Participants are provided with high strength (6 mg) nicotine pouches with smooth flavor.
  Interventions: Other: 6 mg nicotine pouch; Other: Smooth nicotine pouch
- 0 mg + Wintergreen flavor (Experimental): Participants are provided with zero strength (0 mg) nicotine pouches with wintergreen flavor.
  Interventions: Other: 0 mg nicotine pouch; Other: Wintergreen nicotine pouch
- 3 mg + Wintergreen flavor (Experimental): Participants are provided with medium strength (3 mg) nicotine pouches with wintergreen flavor.
  Interventions: Other: 3 mg nicotine pouch; Other: Wintergreen nicotine pouch
- 6 mg + Wintergreen flavor (Experimental): Participants are provided with high strength (6 mg) nicotine pouches with wintergreen flavor.
  Interventions: Other: 6 mg nicotine pouch; Other: Wintergreen nicotine pouch

INTERVENTIONS:
Other: 0 mg nicotine pouch — Oral nicotine pouches that contain 0 mg of nicotine
  Arms: 0 mg + Smooth flavor; 0 mg + Wintergreen flavor
Other: 3 mg nicotine pouch — Oral nicotine pouches that contain 3 mg of nicotine
  Arms: 3 mg + Smooth flavor; 3 mg + Wintergreen flavor
Other: 6 mg nicotine pouch — Oral nicotine pouches that contain 6 mg of nicotine
  Arms: 6 mg + Smooth flavor; 6 mg + Wintergreen flavor
Other: Smooth nicotine pouch — Non-flavored nicotine pouches that are characterized as smooth.
  Arms: 0 mg + Smooth flavor; 3 mg + Smooth flavor; 6 mg + Smooth flavor
Other: Wintergreen nicotine pouch — Menthol flavored nicotine pouches that are characterized as wintergreen.
  Arms: 0 mg + Wintergreen flavor; 3 mg + Wintergreen flavor; 6 mg + Wintergreen flavor

SUMMARY:
The purpose of this clinical trial is to understand the health effects of a new oral nicotine pouch, and also to understand if this product can help reduce traditional cigarette smoking. The main aims are:

1. Understand the impact of nicotine pouch use on toxicant exposure biomarkers, and indicators of potential harms to health.
2. Examine the influence of nicotine pouch use on conventional tobacco product use (cigarettes).

Participants will be randomized to one of six nicotine pouch groups (3 nicotine strengths, each with 2 potential flavors) to use over 16 weeks and asked to reduce their cigarette smoking over that time by at least 75% by substituting with the use of the nicotine pouches. Researchers will compare the outcomes of the different nicotine pouch strengths and flavors to each other. Participants will be asked to complete study questionnaires and provide urine, exhaled carbon monoxide, and mouth cell samples, and other health measurements.

DETAILED DESCRIPTION:
Nicotine Pouches represent a rapidly growing category in the U.S. tobacco market, but little is known about their health effects (including addiction) or effects on cigarette smoking. The investigators propose to use a randomized controlled trial methodology to inform FDA on the effects of nicotine pouch use in smokers interested in reducing their smoking but not quitting smoking. The specific aim of this proposal is to recruit a cohort of 330 current daily smokers with an interest in reducing smoking, and to measure a comprehensive battery of behavioral and health indicators at baseline, and over 16 weeks after being randomized to use Nicotine Pouches containing either 0mg, 3mg or 6mg nicotine in "Smooth" or Wintergreen flavors in a randomized double-blind, placebo-controlled trial. The trial will be conducted at two sites: Penn State Hershey and M.D. Anderson in Texas in order to recruit a diverse sample of smokers. This trial therefore addresses the scientific domain of Product Composition and Design (specifically nicotine content and flavor additives). The central hypothesis is that key markers of toxicity and health effects (e.g. urine NNAL, exhaled carbon monoxide [CO], measures of cigarette addiction [e.g. Penn State Cigarette Dependence Index], oxidative stress and oral B(a)P DNA adducts) will be significantly reduced in smokers who are provided high nicotine (6mg) Nicotine Pouches, relative to 0mg pouches. The investigators will also assess the effects of Nicotine Pouch content on Nicotine Pouch addiction, and the effects of pouch nicotine dose on cigarette and other tobacco product consumption. Lastly, investigators will also compare the effects in those randomized to "Smooth" versus Wintergreen flavors. After the 16-week randomized phase, participants will be encouraged to quit smoking and connected to telephone cessation services and then followed-up 4 weeks later (week 20) in order to ascertain whether the nicotine content of the pouches influenced intention and ability to quit smoking. At the completion of this rigorous double-blind randomized trial investigators will have a better understanding of the effects of Nicotine Pouches (and their nicotine content and flavor characteristics) on cigarette consumption and the resulting changes to markers of health risks, oral health and nicotine addiction.

ELIGIBILITY:
Inclusion Criteria:

* Commonly smoke ≥ 5 cigarettes per day (at least 2 days/week) for at least the prior 12 months
* Exhaled CO measurement of ≥ 6 parts per million at baseline
* Must be interested in reducing cigarette consumption by at least 50% and willing to try nicotine pouches
* Able to understand, read and write in English
* Access to e-mail and a smartphone/computer that has reliable internet connection
* Able to understand and give informed consent

Exclusion Criteria:

* Plans to quit smoking within the next 30 days
* Currently pregnant, breastfeeding, or planning to become pregnant in the next 6 months
* Recent (past 3 months) unstable illness that may increase risks of participation or ability to participate fully (e.g. hospitalization for a mental health condition or substance use disorder in prior 6 months, stroke or myocardial infarction in the past year)
* Serious current respiratory diseases (e.g. exacerbations of asthma or chronic obstructive pulmonary disease [COPD], requiring oxygen or oral prednisone), kidney disease (e.g. requiring dialysis), liver disease (e.g cirrhosis), or any medical disorder/medication that may affect participant safety or biomarker data
* Use of a nicotine pouch or other non-cigarette nicotine product (e-cigarette, pipe, cigar, chew, snus, hookah, IQOS) for 5 or more days in the past 28 days
* Use of illegal drugs daily or weekly in the past 3 months
* Use of combustible (smoked) recreational or medical marijuana weekly in the past 3 months (less frequent smoked medical marijuana or use of other forms of medical marijuana are ok)
* Other member of the household currently participating in the study
* Any other condition that in the opinion of the investigator would make it unlikely that the participant could comply with the study protocol

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Concentration of urinary NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol) | Week 16
  Measure of tobacco-specific nitrosamine

SECONDARY OUTCOMES:
Level of carbon monoxide in exhaled breath | Week 16
  Measure of cigarette smoke exposure obtained with an exhaled carbon monoxide monitor
Concentration of urinary cotinine | Week 16
  Measure of nicotine exposure
Penn State Cigarette Dependence Index score | Week 16
  Measure of cigarette dependence via the Penn State Cigarette Dependence Index. Scale range is 0-20. Higher scores indicate more dependence.
Penn State Nicotine Pouch Dependence Index score | Week 16
  Measure of nicotine pouch dependence via the Penn State Nicotine Pouch Dependence Index. Scale range is 0-20. Higher scores indicate more dependence.
Mean number of cigarettes per day | Week 16
  Measure of mean cigarettes smoked per day
Number of cigarette-free days | Randomization (Week 0) - Week 16
  Measure of number of days abstinent from cigarettes (self-reported)
7-day point prevalence cigarette abstinence | Week 16
  Measure of 7-day point prevalence abstinence biochemically validated with exhaled carbon monoxide < 7ppm

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Foulds, PhD, Principal Investigator — Penn State College of Medicine
Locations (2):
- United States (2):
  - Penn State College of Medicine, Hershey, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Researchers not involved in the execution of this proposed study may request de-identified individual participant data (IPD) collected in the study by contacting the principal investigator, Dr. Jonathan Foulds.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the completion of the main outcome analysis proposed in this study
Access Criteria: Requests for de-identified individual participant data and/or study documents will be considered. The requestor must submit a 1-page abstract of their proposed research, including purpose, analytical plan, and dissemination plans. The Leadership Committee of the Penn State Center for Research on Tobacco and Health will review the abstract and decide based on the individual merits. Review criteria and prioritization of projects include potential of the proposed work to advance public health, qualifications of the applicant, the potential for publication, the potential for future funding, and enhancing the scientific, geographic, and demographic diversity of the research portfolio. Following abstract approval, requestors must receive institutional ethics approval or confirmation of exempt status for the proposed research. An executed data use agreement must be completed prior to data distribution.